CLINICAL TRIAL: NCT06040489
Title: Pilot Study: Oral Treatment of American Tegumentary Leishmaniasis (Cutaneous and Mucosal Forms) in the Elderly
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Brasilia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 57768421.0.0000.5558
Record Dates: First submitted 2022-11-28; First posted 2023-09-15 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-08

CONDITIONS: Leishmaniasis; Brazilian; Leishmaniasis, Mucocutaneous
Keywords: Elderly; Miltefosine; Leishmaniasis; Pentoxifylline; Liposomal amphotericin b; Treatment
MeSH Terms: conditions — Leishmaniasis; Leishmaniasis, Mucocutaneous | interventions — miltefosine; Pentoxifylline; liposomal amphotericin B

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Oral Miltefosine and Pentoxifylline for Cutaneous Leishmaniasis (Experimental)
  Interventions: Drug: Miltefosine 50mg; Drug: Pentoxifylline 400mg
- Oral Miltefosine and Pentoxifylline for Mucous Leishmaniasis (Experimental)
  Interventions: Drug: Miltefosine 50mg; Drug: Pentoxifylline 400mg
- Intravenous Liposomal Amphotericin B for Cutaneous Leishmaniasis (Active Comparator)
  Interventions: Drug: Liposomal Amphotericin B
- Intravenous Liposomal Amphotericin B for Mucous Leishmaniasis (Active Comparator)
  Interventions: Drug: Liposomal Amphotericin B

INTERVENTIONS:
Drug: Miltefosine 50mg — Oral Miltefosine 50mg bid
  Arms: Oral Miltefosine and Pentoxifylline for Cutaneous Leishmaniasis; Oral Miltefosine and Pentoxifylline for Mucous Leishmaniasis
Drug: Pentoxifylline 400mg — Oral Pentoxifylline 400mg tid
  Arms: Oral Miltefosine and Pentoxifylline for Cutaneous Leishmaniasis; Oral Miltefosine and Pentoxifylline for Mucous Leishmaniasis
Drug: Liposomal Amphotericin B — Intravenous 25 to 40mg/kg
  Arms: Intravenous Liposomal Amphotericin B for Cutaneous Leishmaniasis; Intravenous Liposomal Amphotericin B for Mucous Leishmaniasis

SUMMARY:
Randomised clinical trial comparing oral miltefosine associated with pentoxifylline to intravenous liposomal amphotericin b for the treatment of cutaneous and mucosal leishmaniasis

ELIGIBILITY:
Inclusion Criteria:

* Active confirmed cutaneous leishmaniasis ou mucosal leishmaniasis
* Use of highly effective contraceptive method and a negative serologic pregnancy test (beta - HCG), if female in fertile phase
* Agree and sing informed consent form

Exclusion Criteria:

* Previous treatment with leishmanicidal drugs in the last 6 months
* Pre-treatment electrocardiographic changes that contraindicate the use of liposomal amphotericin B (QTc greater than 450ms)
* Serum creatinine or urea 1.5 times the upper limit of normal
* Patients with severe or decompensated liver, kidney, heart disease, Diabetes Mellitus
* history of any hypersensitivity reaction to liposomal amphotericin B, miltefosine and/or pentoxifylline
* Pregnant and breastfeeding women
* Patients with Acquired Immunodeficiency Syndrome (AIDS) or other immunodeficiency

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-06-22 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Cure | 90 days after the begin of treatment
  Complete healing of all lesions (cicatrization of ulcers and complete regression of erythema or infiltration)

SECONDARY OUTCOMES:
Adverse effects | 30 days after drug interruption
  Presence laboratorial or clinica changes during treatment that lead to treatment interruption

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario de Brasilia, Brasília, Federal District, Brazil